CLINICAL TRIAL: NCT01823081
Title: Combined Intravitreal Fasudil and Bevacizumab for Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91128
Record Dates: First submitted 2013-03-21; First posted 2013-04-04 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2012-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravitreal bevacizumab (Avastin) (Active Comparator): Dosage: 1.25 mg/0.05 ml Frequency: 3 consecutive injections every 4 weeks
  Interventions: Drug: Intravitreal injection of bevacizumab (Avastin)
- Combined intravitreal fasudil and bevacizumab (Avastin) (Active Comparator): Dosage: bevacizumab 1.25 mg/0.05 ml + fasudil 0.025mg/0.05ml Frequency: 3 consecutive injections every 4 weeks
  Interventions: Drug: Intravitreal injection of fasudil and bevacizumab (Avastin)

INTERVENTIONS:
Drug: Intravitreal injection of bevacizumab (Avastin)
  Arms: Intravitreal bevacizumab (Avastin)
Drug: Intravitreal injection of fasudil and bevacizumab (Avastin) — intravitreal injections of bevacizumab and fasudil are performed at two different sites (superior temporal and inferior temporal quadrants respectively)
  Arms: Combined intravitreal fasudil and bevacizumab (Avastin)

SUMMARY:
Eligible eyes are randomized to two groups. Group A will receive three intravitreal injections of bevacizumab at 4 week intervals. In group B, three intravitreal injections of combined bevacizumab and fasudil will be performed with the same frequency.

Best corrected visual acuity (BCVA) and central macular thickness (CMT) will be evaluated prior to injections and then every 4 weeks for 6 months. Fluorescein angiography will be performed at baseline and at weeks 12 and 24. The two groups will be compared in terms of BCVA and CMT changes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with diabetic macular edema (DME) and:
* Central macula thickness> 250μm
* Visual acuity < 20/40
* No active proliferative diabetic retinopathy
* No history of intravitreal anti-VEGF drug injection or macular laser photocoagulation (MPC) within the past 3 months

Exclusion Criteria:

* History of vitrectomy
* History of cataract surgery within the past 6 months
* History of glaucoma or uveitis
* Presence of any macular disorder other than DME
* Presence of traction on the macula
* Significant media opacity
* Serum creatinine>3mg/ml

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 6 months
  Snellen E-chart
central macular thickness | 6 months
  spectral domain optical coherence tomography (SD OCT)

SECONDARY OUTCOMES:
Status of macular perfusion | 6 months
  Heidelberg fluorescein angiogram (HRA II)
intraocular inflammation | 6 months
  clinical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran, Iran